CLINICAL TRIAL: NCT06545773
Title: Effect of Conservative Root Canal Preparation on Postoperative Pain: A Randomised Clinical Trial
Brief Title: Postoperative Pain After Conservative Root Canal Preparation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Cagla Vardar, Principal Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IstanbulU-1
Record Dates: First submitted 2024-08-01; First posted 2024-08-09 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Periapical Diseases; Periapical Periodontitis; Postoperative Pain; Pulp Necroses; Flare Up, Symptom
Keywords: pain; Nickel Titanium (NiTi); conservative root canal treatment; minimally invasive; flare-up; analgesic
MeSH Terms: conditions — Periapical Diseases; Periapical Periodontitis; Pain, Postoperative; Dental Pulp Necrosis; Symptom Flare Up; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: ProTaper Next Nickel-Titanium File (PTN) (Experimental): Root canals will be prepared using the ProTaper Next (PTN) instrument. Coronal flaring will be performed using ProTaper Next XA (accessory) in 300 rpm speed and 2 Ncm torque settings. (The same speed and torque settings will be used for all PTN instruments). The glide path will be prepared with ProGlider (Dentsply, Maillefer). ProTaper Next X1 (17 .04) and then X2 (25 .06) will be advanced in the apical direction using a brushing motion. If debris is observed in the apical part of X2 removed from the root canal after reaching the working length, the shaping of the root canal will be completed, and X3 (30 .07) will not be used. If no debris is observed in the apical part of X2 and the #25 K-File reaches the working length loosely, shaping will be continued with X3. Shaping with ProTaper Next X3 will be done in the same way as X1 and X2.
  Interventions: Procedure: Root Canal Treatment with ProTaper Next Nickel-Titanium File (PTN)
- Group 2: TruNatomy Nickel-Titanium File (TN) (Experimental): Root canals will be prepared using the TruNatomy (TN) instrument. Coronal flaring will be performed using the Orifice Modifier (20 .08) at a speed of 400 rpm and a torque setting of 1.5 Ncm. (The same speed and torque settings will be used for all TN instruments.) The Orifice Modifier will be advanced up to 3 mm within the root canal. The guide path will be prepared with TruNatomy Glider (17 .02-variable taper).
  The TruNatomy Prime (26 .04) file will be used in the canal by moving it apically back and forth 2-3 times and not exceeding 2-5 mm, using a brushing motion. Before proceeding to the TruNatomy Medium (35 .04) file, the debris accumulated in the apical part of the Prime file will be checked. If there is no debris between the apical flutes of the TruNatomy Prime file, shaping will be continued with the TruNatomy Medium file. Shaping with TruNatomy Medium will be done in the same manner as with TN Prime.
  Interventions: Procedure: Root Canal Treatment withTruNatomy Nickel-Titanium File (TN)

INTERVENTIONS:
Procedure: Root Canal Treatment with ProTaper Next Nickel-Titanium File (PTN) — ProTaper Next (Dentsply Sirona) is a rotational system made of a nickel-titanium alloy called M-Wire. It has a rectangular cross-sectional design; thus, only two sides touch the root canal. Five files are available: X1 17/. 04, X2 25/.06, X3 30/. 07, X4 40/.06, and X5 50/.06. This file aggressively removes the coronal dentine of root canals due to its large taper. PTN nickel-titanium systemis used in root canal treatments to debride and shape the root canals.
  Arms: Group 1: ProTaper Next Nickel-Titanium File (PTN)
Procedure: Root Canal Treatment withTruNatomy Nickel-Titanium File (TN) — TruNatomy (Dentsply Sirona) is a heat-treated nickel-titanium system that consists of an orifice modifier, glide path, and shaping files. The TruNatomy Small, Prime, and Medium files have sizes of 20/.04, 26/.04, and 35/.04, respectively. It has a rectangular cross-section and a regressive taper. Its slim design allows for a conservative preparation of root canals and the preservation of the coronal dentine. TN nickel-titanium system is used in root canal treatments to debride and shape the root canals.
  Arms: Group 2: TruNatomy Nickel-Titanium File (TN)

SUMMARY:
The goal of this clinical trial is to compare the pain experienced by healthy participants after root canal treatment with small versus large root canal sizes.

The main questions it aims to answer are:

1. Do small and large root canal sizes cause different pain levels?
2. What is the number of painkiller pills taken by each participant?
3. Does small root canal size cause severe pain and facial swelling?

The researcher will perform root canal treatment on lower molar teeth. The researcher will ask about the pain level, painkiller pill number, and swelling on the 6th,12th, 24th, 48th, 72nd hours, and 7th day after the treatment.

DETAILED DESCRIPTION:
Root canal shaping is an essential step for root canal treatment. Necrotic tissues, debris, microorganisms, and organic matter should be removed to clean and disinfect the root canals. Previously, this conventional procedure involved removing excessive dentine from root canals, which weakened the tooth's structural integrity. Due to technological advances, excessive dentine removal is not always necessary. Root canals are claimed to be disinfected despite minimal dentine removal. This concept of treatment is called minimally invasive or conservative root canal treatment.

This study compares postoperative pain after conservative and conventional root canal preparation in healthy participants with necrotic mandibular molars.

Participants will be enrolled after clinical and radiographic examination by an independent endodontist and allocated randomly to conventional or conservative root canal treatment groups. After the root canal treatment, the researcher will send the participants an online questionnaire on the 6th,12th, 24th, 48th, and 72nd hours and 7th day and ask them to rate their pain score according to the Numerical Rating System and the number of painkillers they have taken. The flare-up rate will be determined according to the presence of swelling and severe pain.

An experienced endodontist not involved in the research will monitor eligible participants and clinical treatment protocol.

ELIGIBILITY:
Inclusion Criteria:

* mandibular molar tooth
* asymptomatic apical periodontitis
* pulp necrosis
* periapical lesion index 4 (visible and well-defined periapical lesion)
* absence of pretreatment pain

Exclusion Criteria:

* symptomatic apical periodontitis
* preoperative pain
* sinus tract
* pulpitis
* acute apical abscess
* tooth not being in occlusion
* external and internal root resorption
* open apices
* periodontal probing depth of more than 4 mm
* initial apical file larger than 15 and 20 K-File for mesial and distal canals respectively
* chronic illness, analgesic allergy, prior analgesic and antibiotics usage 12 hours and 3 months before treatment, respectively

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 7 days
  Pain after root canal treatment will be assessed via the Numerical Rating System (NRS) at the 6th, 12th, 24th, 48th, and 72nd hours and on the 7th day. In the NRS, pain is evaluated by numbers from 0 to 10. A score of minimum means no pain, and a score of maximum 10 means the worst pain imaginable.

SECONDARY OUTCOMES:
Analgesic intake | 7 days
  Number of painkiller pills will be asked at 6th, 12th, 24th, 48th and 72nd hours and 7th day.
Flare-up | 7 days.
  Presence of Flare-ups will be determined according to swelling and severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Faruk Haznedaroğlu, Study Director — Istanbul University
Locations (1):
- Istanbul University Faculty of Dentistry, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vardar Korkman C, Haznedaroglu F. Comparison of postoperative pain after instrumentation with TruNatomy or ProTaper Next Ni-Ti systems in mandibular molars with asymptomatic apical periodontitis: a randomized clinical trial. BMC Oral Health. 2025 Apr 13;25(1):564. doi: 10.1186/s12903-025-05895-6. PMID 40223067